CLINICAL TRIAL: NCT02691208
Title: Effectiveness of Acupuncture in Rehabilitation of Physical and Functional Disorders of Women Undergoing Breast câncer Surgery
Brief Title: Acupuncture and Breast Cancer Rehabilitation
Acronym: ACUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Gil Facina, doctor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUSaoPaulo PT 2
Record Dates: First submitted 2016-02-11; First posted 2016-02-25 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Pain
Keywords: acupuncture; breast cancer; rehabilitation; pain
MeSH Terms: conditions — Pain; Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I Kinesiotherapy (Experimental): women with pain treated with a predefinided exercises protocol of 30 minutes.
  Interventions: Other: Kinesiotherapy
- Group II Acupuncture (Experimental): women with pain treated with a predefinided exercises protocol of 30 minutes followed by 30 minutes of acupuncture, used in predefined points
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Kinesiotherapy — Standard therapeutic exercise, pre-defined, based on stretching the neck muscles, shoulder girdle and upper limb exercises for ADM lasting 30 minutes.
  Arms: Group I Kinesiotherapy
Other: Acupuncture — Standard therapeutic exercise, pre-defined, based on stretching the neck muscles, shoulder girdle and upper limb exercises for ADM lasting 30 minutes plus 30 minutes of classical acupuncture using predefined points.
  Arms: Group II Acupuncture

SUMMARY:
The patients were divided into two randomized groups with 24 patients per group, which were given weekly treatment for 10 weeks, one group treated with Kinesiotherapy lasting 30 minutes and the other group followed Kinesiotherapy the same protocol for another 30 minutes acupuncture using predefined points.

The patients were assessed at baseline, after five weeks and at the end of 10 weeks. Responded to an evaluation form about their registration and social data. The physical examination included the assessment of shoulder range of motion, shoulder muscle strength, circumference of the upper limbs and the presence of pain. Questionnaires of quality of life, upper limb function and depression.

DETAILED DESCRIPTION:
They were included in this study patients undergoing surgical treatment for breast cancer, radical or conservative, and to produce pain in the region of the shoulder girdle and upper limb, including thoracic and cervical spine after three months of surgery. Patients over the age of 18 years and level of pain ≥ 3 on the Visual Analogue Scale (VAS). patients with bilateral breast surgery were excluded, metastatic disease, vascular disorders and tactile sensitivity, with diabetes mellitus type I and II uncompensated and with lower level of education than four years. The patients were divided into two randomized groups with 24 patients per group, which were given weekly treatment for 10 weeks, one group treated with Kinesiotherapy lasting 30 minutes and the other group followed Kinesiotherapy the same protocol for another 30 minutes acupuncture using predefined points.

The patients were assessed at baseline, after five weeks and at the end of 10 weeks. Responded to an evaluation form about their registration and social data. The physical examination included the assessment of shoulder range of motion, shoulder muscle strength, circumference of the upper limbs and the presence of pain. questionnaires application EORC QLQ C30 BECK and DASH.

ELIGIBILITY:
Inclusion Criteria:

* underwent surgical treatment of breast cancer, radical or conservative,
* pain in scapular girdle, in the thoracic or cervical spine, after three months surgery.
* level of pain ≥ 3 in the Visual Analogue Scale

Exclusion Criteria:

* bilateral breast surgery,
* metastatic disease,
* vascular and tactile sensitivity disorders,
* uncompensated diabetes mellitus type I and II
* lower education level than four years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Result of rehabilitation about pain, Shoulder Range of Motion, lymphedema presence, upper limb function, Depressive symptoms, Quality of life and Muscle strength with kinesioterapy and acupuncture | two years
  1. Presence of pain by Visual Analog Scale of Pain (VAS).
  2. Shoulder Range of Motion (ROM) by active goniometry of flexion movements, extension, adduction, abduction, internal rotation and external rotation
  3. lymphedema presence through top member perimetry.
  4. upper limb function through the DASH questionnaire.
  5. Depressive symptoms through BECK questionnaire.
  6. Quality of life through the EORTC questionnaire.
  7. Muscle strength of flexion, extension, adduction, abduction, internal rotation and shoulder external rotation with the Hand Held Dynamometer 01,163 model of Lafayette Instrument Company.

CONTACTS AND LOCATIONS:
Overall Officials: Gil Facina, PhD, Principal Investigator — BRazil:Research committee - Recruting
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil